CLINICAL TRIAL: NCT05991206
Title: A Real-World Study of Atezolizumab in Combination With Platinum-Based Doublet Chemotherapy as Neoadjuvant Therapy for Resectable Stage II-IIIB Driver Gene-Negative Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Real-World Study of Atezolizumab in Combination With Platinum-Based Doublet Chemotherapy as Neoadjuvant Therapy for Resectable Stage II-IIIB NSCLC
Status: Recruiting | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Other Study IDs: NATAL RWS
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a descriptive observational study, in which data are collected in an epidemiological fashion and prospective. This study does not intend to intervene the current medical practice of the recruited patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years.
* Provision of fully informed consent prior to any study specific procedures.
* Previously untreated, histologically confirmed resectable stage II, IIIA, IIIB (N2) (AJCC stage VIII) NSCLC; cTNM stage can be confirmed by PET-CT or pathological biopsy; resectable stage II non-small cell lung cancer is defined as radical resection as assessed by a qualified thoracic surgeon; resectable is resectable and potentially resectable as defined by the Expert Consensus on Multidisciplinary Diagnosis and Treatment of Stage III Non-small Cell Lung Cancer (2019 version); resectable includes IIIA (N0-1), some single-station mediastinal lymph node metastases with N2 and some T4 (satellite nodules present in adjacent lobes) N1; potentially resectable includes some stage IIIA and IIIB, including single-station N2 mediastinal lymph node short diameter < 3 cm stage IIIA NSCLC, potentially resectable T3 or T4 central tumors; Solid/solid pulmonary nodules, not pure ground-glass opacity (GGO), are strongly recommended for pathological puncture verification.
* According to the RECIST 1.1 standard, the patient must have at least one measurable lesion.

Exclusion Criteria:

* None

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: stage II, IIIA, IIIB (N2) (AJCC stage VIII) NSCLC
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
MPR Rate | 2 years
  Neoadjuvant therapy-induced tumor regression in pathologically residual tumors <10%

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China